CLINICAL TRIAL: NCT04343261
Title: Convalescent Plasma in the Treatment of COVID 19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFH-20-23
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); COVID; Coronavirus
Keywords: SARS-CoV-1, COVID, Coronavirus, convalescent plasma, plasma
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- COVID-19 patients treated with convalescent plasma (Experimental): Severely ill COVID-19 patients treated with convalescent plasma
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — treatment with 2 Units of convalescent plasma

SUMMARY:
The purpose of this study is to collect blood from previously COVID-19 infected persons who have recovered and use it as a treatment for those who are currently sick with a severe or life-threatening COVID-19 infection.

DETAILED DESCRIPTION:
The purpose of this prospective interventional study is to gain clinical experience using convalescent plasma transfusion administered to critically ill patients with COVID-19.

1 To study the efficacy of plasma from patients recovered from COVID-19 infection with a high neutralizing antibody titer (NAT) as treatment for individuals who are critically ill with COVID-19.

2. Determine if the antibodies from convalescent plasma will suppress virus load in critically ill patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* Age > 18 yrs and < 90 yrs
* Must have laboratory confirmed COVID-19
* Must provide informed consent
* Must have severe or immediately life-threatening COVID-19,

Severe disease is defined as:

* dyspnea,
* respiratory frequency ≥ 30/min,
* blood oxygen saturation ≤ 93%,
* partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300
* lung infiltrates > 50% within 24 to 48 hours

Life-threatening disease is defined as:

* respiratory failure,
* septic shock
* multiple organ dysfunction or failure

Exclusion Criteria:

* No gender exclusion
* Age < 18 yrs and > 90 yrs
* COVID-19 negative

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Latha Dulipsingh, MD, Principal Investigator — Saint Francis Hospital and Medical Centerr/Trinity Health Of New England
Locations (1):
- Trinity Health Of New England, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dulipsingh L, Ibrahim D, Schaefer EJ, Crowell R, Diffenderfer MR, Williams K, Lima C, McKenzie J, Cook L, Puff J, Onoroski M, Wakefield DB, Eadie RJ, Kleiboeker SB, Nabors P, Hussain SA. SARS-CoV-2 serology and virology trends in donors and recipients of convalescent plasma. Transfus Apher Sci. 2020 Dec;59(6):102922. doi: 10.1016/j.transci.2020.102922. Epub 2020 Aug 25. PMID 32883593
- [Result] Ibrahim D, Dulipsingh L, Zapatka L, Eadie R, Crowell R, Williams K, Wakefield DB, Cook L, Puff J, Hussain SA. Factors Associated with Good Patient Outcomes Following Convalescent Plasma in COVID-19: A Prospective Phase II Clinical Trial. Infect Dis Ther. 2020 Dec;9(4):913-926. doi: 10.1007/s40121-020-00341-2. Epub 2020 Sep 20. PMID 32951151
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COVID-19 Patients Treated With Convalescent Plasma
Started | 48
Completed | 40
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — received inadequate amount of antibodies | 7

BASELINE CHARACTERISTICS:
Arm/Group | COVID-19 Patients Treated With Convalescent Plasma
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 17
  More than one race | 12
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Mortality within 28 days
Time Frame: Up to 28 days
Population: 48 patients with severe or life threatening disease with laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection enrolled in the study. 7 patients were excluded from analysis due to receiving plasma with insufficient antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Patients Treated With Convalescent Plasma
Number analyzed (Participants) | 41
Participants | 19

2. Primary Outcome: Viral Load
Description: Median Viral Load at Day 0, Day 3, Day 5, and Day 7 Plasma Viral Load was measured using a research-use only real-time reverse transcription polymerase chain reaction (rRT -PCR) method which targets two regions of the SARS-CoV-2 N gene using TaqMan chemistry.
  The limit of detection for this assay is 75 copies/mL (standard curve of 75 copies/mL to 10,000,000 copies/mL of in vitro transcribed RNA prepared from the full SARS-CoV-2 N gene).
Time Frame: Day 0, Day 3, Day 5, and Day 7
Population: Plasma viral load data was available for 35 out of 41 convalescent plasma recipients on day 0. 22 patients out of 35 had non-detectable levels at Day 0; 25 patients out of 34 had non-detectable levels on Day 3; 20 patients out of 27 had non-detectable levels on Day 5; 20 patients out of 24 had non-detectable levels on Day 7.
Measure: Median (Full Range); unit: copies per mL
Arm/Group | COVID-19 Patients Treated With Convalescent Plasma
Number analyzed (Participants) | 35
copies per mL
  Detectable Viral Load Day 0: number analyzed (Participants) | 13
  Detectable Viral Load Day 0 | 3524 [868 to 8315]
  Detectable Viral Load Day 3: number analyzed (Participants) | 9
  Detectable Viral Load Day 3 | 2033 [243 to 6386]
  Detectable Viral Load Day 5: number analyzed (Participants) | 7
  Detectable Viral Load Day 5 | 315 [214 to 4162]
  Detectable Viral Load Day 7: number analyzed (Participants) | 4
  Detectable Viral Load Day 7 | 494 [102 to 1292]

3. Primary Outcome: Serum Antibody Titers
Description: Median Serum Antibody Titers at Day 0, Day 3, Day 5 and Day 7 Serum Antibody titers were measured using chemiluminescent SARS-CoV-2 immunoglobulin G (IgG) assay from Diazyme (Poway, CA) Positive IgG serum value is > or = 1.0 arbitrary units/mL [AU/mL] (linear reportable range for IgG is 0.20 - 100.00 AU/mL)
Time Frame: Day 0, Day 3, Day 5, and Day 7
Population: 39 out of 41 patients had blood collected on day 0 (pre-transfusion), and on post-transfusion day 3 (n=36), 5 (n=30), and 7 (n=24) and serum antibody titers was assessed at each time point.
Measure: Median (Full Range); unit: arbitrary units/mL (AU/mL)
Arm/Group | COVID-19 Patients Treated With Convalescent Plasma
Number analyzed (Participants) | 39
arbitrary units/mL (AU/mL)
  SARS-CoV-2 Antibodies Day 0 | 18.5 [1.0 to 75.0]
  SARS-CoV-2 Antibodies Day 3: number analyzed (Participants) | 36
  SARS-CoV-2 Antibodies Day 3 | 37.2 [4.5 to 74.6]
  SARS-CoV-2 Antibodies Day 5: number analyzed (Participants) | 30
  SARS-CoV-2 Antibodies Day 5 | 47.4 [6.7 to 80.7]
  SARS-CoV-2 Antibodies Day 7: number analyzed (Participants) | 24
  SARS-CoV-2 Antibodies Day 7 | 55.2 [10.3 to 96.9]

ADVERSE EVENTS:
Time Frame: Treatment and non-treatment related events were collected by non-systematic methods until discharge from the hospital or death, up to 28 days (which ever came first).
Description: Adverse event and/or serious adverse event related to treatment with convalescent plasma
Arm/Group | COVID-19 Patients Treated With Convalescent Plasma
All-Cause Mortality (participants affected / at risk) | 22/48
Serious Adverse Events (participants affected / at risk) | 8/48
Other Adverse Events (participants affected / at risk) | 8/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVID-19 Patients Treated With Convalescent Plasma (N=48)
Persistent Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One subject had persistent hypoxemia and needed extracorporeal membrane oxygenation (ECMO).
Gastrointestinal bleed (Gastrointestinal disorders) | 2 (2) — Two subjects had coffee ground emesis
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — One subject developed acute kidney injury
Atrial fibrillation (Cardiac disorders) | 1 (1) — One subject developed atrial fibrillation
Hypotension; Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One subject became hypotensive, hypoxic and was subsequently intubated
pneumothorax; subcutaneous emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One subject developed pneumothorax and needed a chest tube
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) — One subject had pneumatosis coli of the right colon, air in the superior mesenteric vein and portal venous gas in the liver
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVID-19 Patients Treated With Convalescent Plasma (N=48)
Fever (Immune system disorders) | 1 (1) — Patient developed a fever 1 hour after plasma transfusion
Insufficient Antibodies (Product Issues) | 7 (7) — Patient received convalescent plasma with insufficient antibodies

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT04343261/Prot_SAP_000.pdf
  • Informed Consent Form: Donor Consent (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT04343261/ICF_001.pdf
  • Informed Consent Form: Patient Consent (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT04343261/ICF_002.pdf